CLINICAL TRIAL: NCT06100393
Title: A Feasibility, Prospective, Repeated-measures Investigation of Hearing Outcomes With New Pre-processing Speech Enhancement Algorithms Compared to Standard-of-care Algorithms in Adult Cochlear Implant Recipients: a Master Umbrella Investigation
Brief Title: New Algorithms to Signal Processing for Speech Enhancement in Adult Cochlear Implant Recipients.
Acronym: PRESENCE-MU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AI5842
Record Dates: First submitted 2023-10-02; First posted 2023-10-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Masking Description: Order of IMD and comparator is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub A) (Other)
  Interventions: Device: Investigational Pre-Processing Algorithm (Sub A); Device: Cochlear Limited standard-of-care pre-processing algorithms
- Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub B) (Other): Using Spatial Automation Profile
  Interventions: Device: Cochlear Limited standard-of-care pre-processing algorithms; Device: Investigational Pre-Processing Algorithm (Sub B)
- Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub D) (Other)
  Interventions: Device: Investigational pre-processing algorithm (Sub D); Device: Cochlear Limited standard-of-care pre-processing algorithms
- Other: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub C) (Other): Using Spatial Automation Profile and DNR technology
  Interventions: Device: Cochlear Limited standard-of-care pre-processing algorithms; Device: Investigational Pre-Processing Algorithm (Sub C)

INTERVENTIONS:
Device: Investigational Pre-Processing Algorithm (Sub A) — The algorithms act upon the digital audio signal received by the microphones and other sensors to enhance speech and attenuate noise prior to encoding the signal for delivery to a cochlear implant via the specified system.
  Arms: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub A)
Device: Cochlear Limited standard-of-care pre-processing algorithms — Automatic Gain Control, SNR-NR, Forward Focus
  Arms: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub A); Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub B); Other: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub C)
Device: Investigational Pre-Processing Algorithm (Sub B) — Spatial Automation profile
  Arms: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub B)
Device: Investigational pre-processing algorithm (Sub D) — Microphone miscalibration profile with applied correction method
  Arms: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub D)
Device: Cochlear Limited standard-of-care pre-processing algorithms — Standard microphone calibration profile
  Arms: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub D)
Device: Investigational Pre-Processing Algorithm (Sub C) — Spatial Automation profile and DNR algorithm
  Arms: Other: Investigational pre-processing algorithm/Standard of Care pre-processing algorithm (Sub C)

SUMMARY:
The purpose of this clinical investigation is to develop pre-processing strategies to enhance speech and reduce noise for CI listeners. The Master Umbrella Clinical Investigation will be comprised of several sub-investigations, which will aim to optimize speech enhancement algorithms, to improve real-world functionality, and to incorporate them efficiently into CI speech processors.

DETAILED DESCRIPTION:
This is a feasibility, prospective, multi-center, single-subject, repeated-measures clinical investigation in experienced adult cochlear implant users. The Master Umbrella design will enable the execution of a series of sub-investigations in the same user population, with the goal to evaluate a range of speech enhancement pre-processing algorithms in separate sub-investigations. The primary objectives for each sub-investigation will be consistent with the master umbrella investigation, with secondary and exploratory objectives selected based on the algorithm to be investigated. Secondary and exploratory objectives will be described in the sub-investigation documentation.

ELIGIBILITY:
Inclusion Criteria:

* User of an approved Nucleus cochlear implant.
* User of the ACE (Advanced Combination Encoder) sound processing strategy.
* Aged 18 years or older (no upper age limit).
* Able to score 20% or more at +10 dB SNR or have an adaptive Speech Recognition Threshold (SRT) of 12 dB or less CI alone on a sentence in babble test.*
* Fluent speaker in the language used to assess speech perception performance, as determined by the investigator.
* Willing and able to provide written informed consent.
* ≥3 months post cochlear implant activation

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Additional health factors, known to the investigator, that would prevent or restrict participation in the audiological evaluations.
* Investigator site personnel directly affiliated with this study and/or the investigator's immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Australian Sentence Test in Noise (AuSTIN) | 1 day - Immediately post-screening
  To determine whether the research algorithm provides non-inferior performance to the standard-of-care algorithm for sentences in noise using an adaptive sentence test in noise scores.
  Scoring: AuSTIN is scored as a Speech Reception Threshold (SRT), which reflects the volume of speech signal (in decibels, dB) relative to the background noise required for the subject to achieve 50% correct. For example, a score of 2dB SRT means the subject requires the speech to be 2dB louder than the background noise in order to correctly identify 50% of the target sentence.
  Range: -30dB to +30dB. Lower scores reflect a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Cochlear Melbourne, Melbourne, Victoria
  - HEARnet Clinical Studies, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No